CLINICAL TRIAL: NCT00140920
Title: A Study to Compare Pre-Operative Administration of Rofecoxib Vs Post-Operative Administration of Diclofenac or Rofecoxib in the Treatment of Post-Operative Pain After Total Knee Joint Replacement in Patients With Osteoarthritis of the Knee.
Brief Title: A Study of Rofecoxib in the Treatment of Post-Operative Pain After Total Knee Joint Replacement (0966-259)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment/study discontinued after withdrawal of marketing authorisation. No data entered.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0966-259; 2005_054
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — rofecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0966; rofecoxib
Drug: Comparator: diclofenac 2x 75 mg

SUMMARY:
A study to compare pre-operative administration of rofecoxib versus post-operative administration of diclofenac or rofecoxib, respectively, in the treatment of post-operative pain after total knee joint replacement in patients with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Males or females at least 18 years of age who have osteoarthritis of the knee and have undergone total knee joint replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2004-05-25 (Actual); Primary Completion 2004-09-27 (Actual); Study Completion 2004-09-27 (Actual)

PRIMARY OUTCOMES:
Quantity of patient controlled
Post-operative morphine administration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html